CLINICAL TRIAL: NCT01058876
Title: Nicotine Regulation/Response to Low Yield Cigarettes in African-Americans vs. Whites
Brief Title: Comparison of Low Yield Cigarettes in African Americans vs. Whites
Acronym: 6162-AAPK2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10-00158; NIDA DA002277 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Cigarette Smoking
Keywords: Smoking; nicotine
MeSH Terms: conditions — Cigarette Smoking; Smoking | interventions — Cotinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Cigarette (Experimental): African American and White Smokers will smoke their usual cigarette and also undergo an oral pharmacokinetics protocol after administration of 3 mg deuteriumlabeled nicotine and 5 mg deuterium-labeled cotinine.
  Interventions: Drug: Deuterated nicotine and cotinine
- Low-yield Cigarette (Experimental): African American and White smokers will smoke a commercial cigarette with a machine-determined nicotine yield of approximately 50% of their "usual" brand.
  Interventions: Drug: Deuterated nicotine and cotinine

INTERVENTIONS:
Drug: Deuterated nicotine and cotinine — used as a marker for pharmacokinetic studies

SUMMARY:
The investigators' general hypothesis is that African-Americans (AAs) smoke more for positive reinforcement from nicotine with a "peak-seeking" pattern of smoking (smoking individual cigarettes more intensively with greater intake of nicotine and tobacco smoke toxins), while whites smoke more for negative reinforcement with a "trough-maintaining" pattern (avoiding withdrawal by maintaining more consistent nicotine levels throughout the day by means of a more regular smoking pattern). We, the investigators, believe that these patterns are linked to identifiable racial differences in nicotine pharmacology.

For this study we hypothesize that if AAs behave more like nicotine "peak-seeker" while whites behave more like nicotine "trough-maintainers", that AAs will respond to switching from regular to low nicotine yield commercial cigarettes by smoking each cigarette relatively more intensively with a relatively smaller increase in daily cigarette consumption (cigarettes per day or CPD) as compared to whites.

DETAILED DESCRIPTION:
Several lines of evidence indicate that AAs are more highly addicted to cigarette smoking than are whites. AAs are more likely to smoke their first cigarette within 10 minutes of awakening, an indicator of the severity of the dependence. They are more likely to want to quit smoking and are more likely to try to quit (attempts lasting at least 24 hours, but are significantly less likely than whites to be successful abstainers at one year. The quit ratio (former smokers/ever smokers) was recently reported to be 37.3% in AAs compared to 51% for whites (2).

NICOTINE REGULATION IN AAS AND WHITES: In general smokers regulate (titrate) their smoking to take in about the same amount of nicotine from day to day. This behavior is well demonstrated in studies of smokers smoking commercial cigarettes of differing yields, showing that smokers take in similar amounts of nicotine from high- and low-yield cigarettes. NCI MONOGRAPH 13 summarized the data on nicotine and low yield cigarettes and concluded that low yield cigarettes presented the same health risks as high yield cigarettes (12). However, most or all of the research on nicotine titration appears to have been done primarily in white smokers.

We believe that nicotine titration patterns will differ in AAs compared to whites, based on the hypothesis that AAs smoke more for the positive reinforcing effects of individual cigarettes, while whites smoke more to maintain a consistent level of nicotine. We predict that the response to switching from regular to low yield cigarettes in AAs will differ in that they will try to take in more nicotine per cigarette by smoking more intensively, but will be less likely to try to regulate their total daily intake of nicotine compared to whites.

Melanin: A recent study (14) showed that levels of facultative melanin (includes both genetically and exposure influenced melanin) in the skin are significantly and positively related to cigarettes per day, the Fagerstrom score, and cotinine levels. By measuring melanin levels in our own study subjects, we will be able to determine if there is a relationship between melanin levels and nicotine pharmacokinetics.

This is a non-randomized, non-blinded, two treatment arm crossover study with an oral nicotine and cotinine pharmacokinetic study. Cigarettes will be supplied for both treatment arms and subjects will smoke ad libitum. During the first arm, the subject will smoke their "usual" cigarettes and also undergo an oral pharmacokinetics protocol. During the second arm, subjects will smoke a commercial cigarette with a machine-determined nicotine yield of approximately 50% of their "usual" brand.

Blood and urine samples will be collected throughout the study and analyzed by our usual methods.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female (balanced numbers)
* Age: 18- 65
* Race/ethnicity: African-American or White (based on two parents who self- identify as AA or White, respectively)
* Smoking Status: Current daily smoker of at least 10 cigarettes per day; either menthol or non-menthol. Screening saliva cotinine level of > 100 ng/ml.

Healthy by history and assessment of vital signs.

Exclusion Criteria:

* Evidence of cardiac disease by history
* Recent or current history of asthma or severe allergic rhinitis
* Hypertension (blood pressure [BP] >140/90 at screening after 5 min rest)
* Serious medical or psychiatric condition or other condition requiring regular medication use
* Lack of access to a refrigerator to store saliva specimens collected at home
* Morbid obesity (body mass index [BMI]>35)
* Current illicit drug use by history and tox screen (however subjects using marijuana may be included if they are not daily users and will agree to abstain from the time of screening until the end of the study)
* Pregnancy or breastfeeding
* Significant history of fainting, "bad veins", discomfort with blood draws
* Current or recent alcohol or drug abuse
* Inability to speak English/read forms or aversion to filling out forms
* Multiple or unexplained "no shows" for screening/study visits or other noncompliance with study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Nicotine clearance | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Neal L Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco General Hospital, San Francisco, California, United States